CLINICAL TRIAL: NCT07145294
Title: Induced Pluripotent Stem Cells-derived Small Extracellular Vesicles May Promote Neurological Function and Improve Cognitive Impairment in Acute Ischemic Stroke Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hongmei Wang (Other)
Responsible Party: Sponsor-Investigator, Hongmei Wang, Chief Physician of the Department of Neurology, Shanghai Sixth People's Hospital, and Youth Council Member of the Chinese Stroke Association, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-100-（1）
Record Dates: First submitted 2025-08-10; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment
Keywords: Neuronal damage and cognitive dysfunction induced by acute cerebral ischemia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSCI+iEV (Experimental): Intranasal administration of iEV, twice a week, 2 ml each time (at a concentration of 2×10¹⁰/ml), for 12 consecutive weeks.
  Interventions: Biological: iEV; Other: Basic treatments
- PSCI+Control (Placebo Comparator): Control
  Interventions: Other: Basic treatments

INTERVENTIONS:
Biological: iEV — Intranasal administration of iEV, twice a week, 2 ml each time (at a concentration of 2×10¹⁰/ml), for 12 consecutive weeks.
  Arms: PSCI+iEV
Other: Basic treatments — Basic treatments for cerebrovascular diseases such as antiplatelet aggregation, blood pressure control, blood glucose control, blood lipid control, and plaque stabilization.

SUMMARY:
This study primarily evaluates whether iEV nasal administration can improve neurological impairment and cognitive dysfunction in patients with acute cerebral infarction and cognitive impairment, and preliminarily explores its clinical efficacy.

DETAILED DESCRIPTION:
1. It is planned to enroll 40 patients with post - stroke cognitive impairment (PSCI, i.e., acute ischemic stroke (AIS) combined with cognitive impairment) who are hospitalized in the Department of Neurology and Stroke Ward of Shanghai Sixth People's Hospital. These patients should have had an AIS onset within 14 days. They will be divided into the PSCI + treatment group and the PSCI + control group according to a random number table, with 20 patients in each group.
2. Enrolled patients need to first complete blood tests such as blood routine and blood biochemistry, as well as skull MRI or skull CT examinations. The total course of treatment for both groups will be 12 weeks.
3. Both the treatment group and the control group will receive conventional basic treatment for cerebrovascular diseases. In addition, the treatment group will be given intranasal iEV administration, twice a week, 2 ml each time (with a concentration of 2×10¹⁰/ml), for 12 consecutive weeks. Before treatment and 12 weeks after treatment, the severity of neurological impairment, self - care ability, disability status, and cognitive function status will be evaluated to assess the therapeutic effect of iEV on neurological impairment and cognitive dysfunction in PSCI patients.
4. Before intranasal iEV treatment and 12 weeks after treatment, blood samples will be collected respectively to detect changes in indicators such as nerve cell damage, pro - inflammatory factors, angiogenesis, and blood - brain barrier disruption, so as to clarify the neuroprotective mechanism of iEV in PSCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Diagnosed with acute ischemic stroke (AIS) according to WHO criteria.
* Time from onset to enrollment ≤ 2 weeks (stable condition after admission and able to cooperate with cognitive assessment), accompanied by manifestations of cognitive impairment, with a score of < 26 on the Montreal Cognitive Assessment (MoCA) scale.
* Cerebral MRI or CT scan shows stroke lesions related to the condition.
* Subjects or their family members voluntarily participate and sign the informed consent form.

Exclusion Criteria:

* A diagnosis of cognitive impairment prior to the onset of AIS;
* Presence of aphasia, hearing impairment, visual impairment, dysarthria, or other conditions that prevent completion of neuropsychological assessments;
* Patients with mental illnesses such as depression, anxiety disorder, or schizophrenia;
* Patients with severe diseases of the heart, liver, lungs, kidneys, or other vital organs;
* Patients with disturbed consciousness, a history of long-term alcohol consumption, a history of severe head trauma, or those who cannot cooperate with cognitive function tests for various reasons;
* illiterate patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
NIHSS | From enrollment to the end of treatment at 12 weeks
  The **National Institutes of Health Stroke Scale (NIHSS)** is a standardized, 11-item assessment tool used to quantify the severity of neurological deficits in patients with acute stroke. Designed to provide objective measurements, it evaluates key domains including level of consciousness (alertness, orientation, and ability to follow commands), gaze, visual fields, facial palsy, motor strength in arms and legs, limb ataxia, sensory function, language (ability to comprehend and express), dysarthria (speech clarity), and extinction/inattention (neglect of sensory or motor stimuli). Each item is scored from 0 (no deficit) to a maximum of 2, 3, or 4 points, depending on the domain, with total scores ranging from 0 (no neurological impairment) to 42 (severe impairment). Widely used in clinical practice, emergency care, and research, the NIHSS helps guide treatment decisions (such as eligibility for thrombolysis or thrombectomy), track neurological changes over time, and predict patient ou
mRS | From enrollment to the end of treatment at 12 weeks
  The **Modified Rankin Scale (mRS)** is a widely used, standardized tool to assess functional outcome and disability in patients following neurological events, most commonly stroke. Ranging from 0 to 6, it categorizes a patient's level of independence in daily activities based on their ability to perform tasks without assistance. A score of 0 indicates no symptoms or disability, while 1 reflects minor symptoms with no functional impairment. Scores of 2 and 3 denote mild to moderate disability, where patients require some help but can walk unassisted (2) or need significant assistance and may have difficulty walking (3). A score of 4 indicates severe disability, with patients unable to walk or attend to their own bodily needs without constant care. A score of 5 represents complete dependence on others for all aspects of daily living, and 6 signifies death. The mRS is valued for its simplicity, clinical relevance, and ability to track recovery over time, making it essential for guiding p
ADL | From enrollment to the end of treatment at 12 weeks
  The **Activities of Daily Living (ADL) scale** is a standardized assessment tool used to evaluate an individual's ability to perform essential self-care and daily tasks independently. Focused on functional capacity, it typically includes key activities such as bathing, dressing, grooming, toileting, feeding, transferring (e.g., moving from bed to chair), and maintaining continence. Scoring systems vary slightly across versions (e.g., Barthel Index, Katz Index), but most rate each activity on a scale reflecting independence (e.g., "able to perform without help") to dependence (e.g., "requires full assistance" or "unable to perform"). Total scores quantify the level of functional impairment, with higher scores indicating greater independence and lower scores signaling increased reliance on others. Widely used in healthcare settings-particularly for patients with stroke, dementia, or chronic illness-the ADL scale helps guide care planning, assess recovery progress, determine long-term ca
MoCA | From enrollment to the end of treatment at 12 weeks
  The **Montreal Cognitive Assessment (MoCA)** is a brief, standardized tool designed to screen for mild cognitive impairment and detect early signs of cognitive decline, often used in clinical settings to evaluate individuals at risk for conditions like Alzheimer's disease or vascular dementia. Comprising 30 points across multiple cognitive domains, it assesses attention and concentration, executive functions (e.g., planning, problem-solving), memory (immediate and delayed recall), language (naming, fluency, comprehension), visuospatial abilities (e.g., copying a complex figure), calculation, and orientation to time and place. Each task is scored based on performance, with points deducted for errors or incomplete responses. A total score of 26 or higher is generally considered normal, while scores below 26 indicate varying degrees of cognitive impairment, with lower scores reflecting more significant deficits. Valued for its sensitivity to mild impairments-often missed by simpler tools
MMSE | From enrollment to the end of treatment at 12 weeks
  The **Mini-Mental State Examination (MMSE)** is a widely used, brief screening tool designed to assess global cognitive function, primarily to detect cognitive impairment or dementia. Consisting of 30 points, it evaluates key cognitive domains including orientation to time and place (e.g., identifying the current date, season, or location), registration (remembering a list of words), attention and calculation (e.g., serial subtraction or spelling backward), recall (retrieving the earlier list of words), language (naming objects, following commands, writing a sentence, or copying a design), and comprehension. Each task is scored based on accuracy or completion, with points awarded for correct responses. A total score of 27-30 is typically considered within the normal range, 21-26 indicates mild impairment, 10-20 reflects moderate impairment, and scores below 10 signify severe cognitive decline. While valued for its simplicity and widespread use in clinical and research settings, the MM

SECONDARY OUTCOMES:
Indicators of pro-inflammatory factors | From enrollment to the end of treatment at 12 weeks
  Changes in indicators of pro-inflammatory factors (including IL-6, IL-1β, TGF-β).
Indicators of blood-brain barrier disruption | From enrollment to the end of treatment at 12 weeks
  Changes in indicators of blood-brain barrier disruption(VE-cadherin、Claudin-5、ZO-1).
Indicators of neuronal injury | From enrollment to the end of treatment at 12 weeks
  Changes in indicators of neuronal injury (NSE, S100β, TDP-43, BDNF, GFAP).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No